CLINICAL TRIAL: NCT00982865
Title: A Multicenter, Open Label, Phase I Trial of the MEK Inhibitor MSC1936369B Given Orally to Subjects With Solid Tumours
Brief Title: Trial of MSC1936369B in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28062; 2007-004665-18 (EudraCT Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors; Cancer
Keywords: MEK inhibitor; Cancer; Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MSC1936369B Regimen 1 (Experimental): Subjects will be administered MSC1936369B (pimasertib) capsules 1 to 120 milligram (mg) orally, once daily (QD) on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until progressive disease (PD) or intolerable toxicity or investigator/subject decision.
  Interventions: Drug: MSC1936369B
- MSC1936369B Regimen 2 (Experimental): MSC1936369B Regimen 2 (Without Food Effect): Subjects will be administered MSC1936369B capsules 1 to 255 mg orally QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
  MSC1936369B Regimen 2 (With Food Effect): : Subjects will be administered MSC1936369B capsules 90 or 150 mg orally QD on Day 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision. Subjects in the Regimen 2 FE cohort were assigned in a 1:1 ratio to either the fed/fasted sequence or fasted/fed sequence for Day 1 of Cycle 1 and Day 1 of Cycle 2.
  Interventions: Drug: MSC1936369B
- MSC1936369B Regimen 3 once daily (Experimental): Subjects will be administered MSC1936369B capsules 60 to 90 mg orally QD in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
  Interventions: Drug: MSC1936369B
- MSC1936369B Regimen 3 twice daily (BID) (Experimental): Subjects will be administered MSC1936369B capsules 45 to 75 mg orally BID in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
  Interventions: Drug: MSC1936369B

INTERVENTIONS:
Drug: MSC1936369B
  Other Names: Pimasertib
  Arms: MSC1936369B Regimen 1
Drug: MSC1936369B
  Other Names: Pimasertib
  Arms: MSC1936369B Regimen 2
Drug: MSC1936369B
  Other Names: Pimasertib
  Arms: MSC1936369B Regimen 3 once daily
Drug: MSC1936369B
  Other Names: Pimasertib
  Arms: MSC1936369B Regimen 3 twice daily (BID)

SUMMARY:
This is a first in man trial with a primary objective being the determination of the Maximum Tolerated dose (MTD) and the dose-limiting toxicity (DLT) in several regimens of MEK inhibitor MSC1936369B administered orally once a day, in subjects with malignant solid tumors to see how safe is treatment with MSC1936369B.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed solid tumor which is locally advanced or metastatic, and either refractory after standard therapy for the disease or for which no effective standard therapy is available. In the regimen 3, regimen 2 food-effect, and BID cohorts, the tumor type will be restricted to melanoma.
* Age greater than or equal to (>=) 18 years
* Has read and understands the informed consent form and is willing and able to give informed consent. Fully understands requirements of the trial and willing to comply with all trial visits and assessments

Exclusion Criteria:

* Bone marrow impairment as evidenced by Haemoglobin less than (<) 9.0 gram per deciliter (g/dL), Neutrophil count < 1.0*10^9/Liter, platelets < 100*10^9/Liter
* Renal impairment as evidenced by serum creatinine > 1.5*upper limit normal (ULN), and/or calculated creatinine clearance < 60 milliliter per minute (mL/min)
* Liver function abnormality as defined by total bilirubin > 1.5*ULN, or aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5*ULN, for subjects with liver involvement AST/ALT > 5*ULN
* INR > 1.5*ULN
* Serum calcium > 1*ULN
* History of central nervous system (CNS) metastases, unless subject has been previously treated for CNS metastases, is stable by computer tomography (CT) scan without evidence of cerebral oedema, and has no requirements for corticosteroids or anticonvulsants
* History of difficulty swallowing, malabsorption or other chronic gastro-intestinal disease or conditions that may hamper compliance and/or absorption of the tested product
* Eastern Cooperative Oncology Group Performance status (ECOG PS) greater than (>) 1
* Known human immunodeficiency virus (HIV) positivity, active hepatitis C, or active hepatitis B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2007-12-31 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (9):
- Westmead Hospital, Westmead, Australia
- Belgium (2):
  - Jules Bordet Institute, Brussels
  - Ghent University Hospital, Ghent
- France (5):
  - Institute Bergonié, Bordeaux
  - Hôpital Beaujon, Paris
  - Hopital Saint Louis, Paris
  - Centre Eugène Marquis, Rennes
  - Institute Claudius Regaud, Toulouse
- Netherlands Cancer Institute - Antonie van Leeuwenhoek Hospital, Amsterdam, Netherlands

REFERENCES:
- [Derived] Lebbe C, Italiano A, Houede N, Awada A, Aftimos P, Lesimple T, Dinulescu M, Schellens JHM, Leijen S, Rottey S, Kruse V, Kefford R, Raymond E, Faivre S, Pages C, Gomez-Roca C, Schueler A, Goodstal S, Massimini G, Delord JP. Selective Oral MEK1/2 Inhibitor Pimasertib in Metastatic Melanoma: Antitumor Activity in a Phase I, Dose-Escalation Trial. Target Oncol. 2021 Jan;16(1):47-57. doi: 10.1007/s11523-020-00767-1. PMID 33211315
- [Derived] Delord JP, Italiano A, Awada A, Aftimos P, Houede N, Lebbe C, Pages C, Lesimple T, Dinulescu M, Schellens JHM, Leijen S, Rottey S, Kruse V, Kefford R, Faivre S, Gomez-Roca C, Scheuler A, Massimini G, Raymond E. Selective Oral MEK1/2 Inhibitor Pimasertib: A Phase I Trial in Patients with Advanced Solid Tumors. Target Oncol. 2021 Jan;16(1):37-46. doi: 10.1007/s11523-020-00768-0. PMID 33170484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): December 2007/March 2012. Last subject completed: April 2016.
Pre-assignment Details: A total of 182 subjects entered the trial, of which 2 did not receive any treatment. 180 subjects received the study treatment and were included in the subject disposition table.
Groups:
- MSC1936369B Regimen 1: Subjects received MSC1936369B capsules 1 to 120 mg orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B Regimen 2 (Without Food Effect + With Food Effect): MSC1936369B Regimen 2 (Without Food Effect): Subjects received MSC1936369B capsules 1 to 255 mg orally QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision. MSC1936369B Regimen 2 (With Food Effect): Subjects received MSC1936369B capsules 90 or 150 mg orally QD on Day 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision. Subjects in the Regimen 2 FE cohort were assigned in a 1:1 ratio to either the fed/fasted sequence or fasted/fed sequence for Day 1 of Cycle 1 and Day 1 of Cycle 2.
- MSC1936369B Regimen 3 Once Daily (QD): Subjects received MSC1936369B capsules 60 to 90 mg orally QD in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B Regimen 3 Twice Daily (BID): Subjects received MSC1936369B capsules 45 to 75 mg orally BID in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Period: Overall Study
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily (BID)
Started | 49 | 82 | 15 | 34
Completed | 49 | 82 | 15 | 34
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least 1 dose of MSC1936369B treatment.
Groups:
- MSC1936369B Regimen 3 Twice Daily: Subjects received MSC1936369B capsules 45 to 75 mg orally BID in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- Total: Total of all reporting groups
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily | Total
Number analyzed (Participants) | 49 | 82 | 15 | 34 | 180
Age, Customized [Number; unit: Participants]
  >= 18 - <45 Years | 4 | 10 | 4 | 7 | 25
  >=45 - <65 Years | 30 | 49 | 9 | 13 | 101
  >=65 Years | 15 | 23 | 2 | 14 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 9 | 11 | 70
  Male | 29 | 52 | 6 | 23 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experienced Any Dose-Limiting Toxicity (DLT) Over the First Cycle - Day 1 to 21
Description: DLT was defined as any of following toxicities at any dose level according to using National Cancer Institute Common Terminology Criteria for Adverse Events (AEs) v3.0(CTCAE), probably or possibly related to trial medication by investigator or sponsor: a)Any Grade 3 or more non-haematological toxicity excluding: (i)Grade 3 asymptomatic increase in liver function tests (Aspartate Aminotransferase, Alanine transaminase, Alkaline Phosphatase reversible within 7 days for subjects without liver involvement, or grade 4 for subjects with liver involvement; (ii)Grade 3 vomiting if it is encountered despite adequate and optimal therapy (e.g. serotonin [5HT3] antagonists and corticosteroids); (iii)Grade 3 diarrhoea if it is encountered despite adequate and optimal anti diarrhoea therapy; b)Grade 4 neutropenia of >5 days duration or febrile neutropenia lasting for more than 1 day; c)Grade 4 thrombocytopenia >1 day or grade 3 with bleeding; d)Any treatment delay >2 weeks due to drug-related AEs.
Time Frame: Day 1 up to Day 21 of Cycle 1
Population: Dose Escalation Analysis Set included all subjects who meet at least 1 of following criteria:
  subjects who experienced any DLT during Cycle 1 & who received planned treatment.
Measure: Number; unit: Subjects
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily
Number analyzed (Participants) | 44 | 74 | 15 | 33
Subjects | 2 | 6 | 0 | 6

2. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAE), Serious TEAEs, TEAEs Leading to Discontinuation
Description: AE was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 253 weeks. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 253 weeks
Population: Safety Analysis Set (SAF) included all subjects who received at least 1 dose of MSC1936369B treatment.
Measure: Number; unit: Subjects
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily
Number analyzed (Participants) | 49 | 82 | 15 | 34
Subjects
  TEAEs | 47 | 82 | 15 | 34
  Serious TEAEs | 23 | 45 | 8 | 21
  TEAEs leading to discontinuation | 13 | 22 | 2 | 6

3. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) Leading to Death
Time Frame: Baseline up to 253 weeks
Population: ALL subject analysis set was used which included all the subjects who signed the informed consent form and entered the study.
Measure: Number; unit: Subjects
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily
Number analyzed (Participants) | 49 | 83 | 15 | 35
Subjects | 10 | 14 | 2 | 2

4. Secondary Outcome: Number of Subjects With Clinical Significant Laboratory Abnormalities and Vital Signs Reported as Treatment Emergent Adverse Events
Description: Any clinically significant changes in laboratory evaluations and vital signs were recorded as treatment emergent adverse events. The clinical laboratory parameters that were assessed included: Hematological parameters, Blood chemistry parameters, Urinalysis and the vital signs that were assessed included: Blood pressure, Heart rate, Temperature and Weight. SAF analysis was used.
Time Frame: Baseline up to 253 weeks
Population: SAF analysis was used.
Measure: Number; unit: Subjects
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily
Number analyzed (Participants) | 49 | 82 | 15 | 34
Subjects
  Haemoglobin decreased | 1 | 2 | 0 | 0
  Anaemia | 10 | 23 | 3 | 3
  Lymphopenia | 3 | 7 | 0 | 0
  Thrombocytopenia | 3 | 6 | 2 | 1
  Platelet count decreased | 0 | 1 | 0 | 0
  Neutropenia | 0 | 4 | 0 | 1
  Leukopenia | 0 | 0 | 1 | 0
  Pancytopenia | 0 | 0 | 0 | 1
  Hyponatraemia | 0 | 1 | 0 | 1
  Hypokalaemia | 4 | 10 | 2 | 2
  Hyperkalaemia | 1 | 0 | 0 | 0
  Hypocalcaemia | 2 | 7 | 0 | 1
  Hypercalcaemia | 0 | 3 | 0 | 0
  Hypomagnesaemia | 2 | 3 | 2 | 0
  Hypophosphataemia | 0 | 2 | 0 | 0
  Hepatic enzyme increased | 0 | 1 | 0 | 0
  Hepatic function abnormal | 0 | 1 | 0 | 0
  Alanine aminotransferase increased | 0 | 1 | 0 | 2
  Aspartate aminotransferase increased | 1 | 1 | 0 | 2
  Blood alkaline phosphatase increased | 1 | 0 | 0 | 1
  Hyperbilirubinaemia | 1 | 1 | 0 | 0
  Blood lactate dehydrogenase increased | 1 | 0 | 0 | 1
  Blood creatine phosphokinase increased | 1 | 2 | 1 | 5
  Blood creatinine increased | 0 | 1 | 0 | 0
  Blood 25-hydroxycholecalciferol decreased | 1 | 1 | 0 | 0
  Vitamin D decreased | 0 | 1 | 0 | 0
  Blood parathyroid hormone increased | 1 | 1 | 0 | 0
  Hyperglycaemia | 0 | 1 | 0 | 0
  C-reactive protein increased | 0 | 1 | 0 | 0
  Proteinuria | 0 | 0 | 1 | 1
  Hyperthyroidism | 0 | 0 | 0 | 1
  Hypoalbuminaemia | 3 | 4 | 0 | 2
  Weight increased | 0 | 3 | 0 | 3
  Weight decreased | 6 | 8 | 4 | 2
  Hyperthermia | 1 | 5 | 0 | 1
  Hypertension | 7 | 5 | 1 | 4
  Hypotension | 3 | 1 | 2 | 0
  Heart rate increased | 1 | 0 | 0 | 0
  Tachycardia | 3 | 0 | 2 | 0
  Blood potassium increased | 1 | 0 | 0 | 0

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MSC1936369B: Regimen 1
Description: Pharmacokinetic (PK) parameter Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours (h) post-dose on Cycle 1(C1) Day 1 (D1), Cycle 1 Day 12 (D12) and Cycle 3 (C3) Day 1
Population: PK analysis set: subjects received at least 1 dose of drug & provided sufficient PK serum samples for at least 1st 24h following 1st dose of C1D1. Number of Participants Analyzed=subjects evaluable for this endpoint & Number analyzed=subjects evaluated at specified time point & "0"indicates no subject analyzed for that specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- MSC1936369B 1 mg: Subjects received 1 mg of MSC1936369B (capsule formulation) orally, once daily on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 1.5 mg: Subjects received 1.5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 2.5 mg: Subjects received 2.5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 3.5 mg: Subjects received 3.5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 7 mg: Subjects received 7 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 14 mg: Subjects received 14 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 28 mg: Subjects received 28 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 45 mg: Subjects received 45 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 68 mg: Subjects received 68 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 94 mg: Subjects received 94 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 120 mg: Subjects received 120 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 4 | 3 | 13
nanogram per milliliter (ng/mL)
  C1D1 | 2.02 (41.0) | 3.20 (45.5) | 4.21 (47.9) | 6.69 (62.9) | 12.60 (15.4) | 62.32 (33.6) | 126.21 (70.2) | 212.96 (106.3) | 357.39 (30.7) | 325.99 (31.8) | 428.85 (57.9)
  C1D12: number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 11
  C1D12 | 2.92 (39.0) | 2.69 (10.1) | 6.29 (40.6) | 9.75 (63.3) | 21.93 (110.5) | 54.47 (116.2) | 150.67 (78.1) | 175.94 (47.5) | 413.58 (9.1) | 602.12 (11.0) | 425.26 (71.0)
  C3D1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 1 | 3 | 2 | 0 | 2 | 7
  C3D1 | 2.00 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.90 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 5.60 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 8.06 (30.3) | 10.90 (68.5) | 51.30 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 84.70 (78.8) | 167.75 (15.5) |  | 282.44 (14.9) | 652.70 (48.3)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MSC1936369B: Regimen 2 (Without Food Effect)
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure and "Number analyzed" signifies those who were evaluated at the specified time point. Data was not available for categories with Number analyzed= 0 as no subject analyzed at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MSC1936369B 2 mg: Subjects received 2 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 3.5 mg: Subjects received 3.5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 5 mg: Subjects received 5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 7 mg: Subjects received 7 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 28 mg: Subjects received 28 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 45 mg: Subjects received 45 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 68 mg: Subjects received 68 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 94 mg: Subjects received 94 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 120 mg: Subjects received 120 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 150 mg: Subjects received 150 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 and Day 2 of 21-day treatment cycle in either fed or fasted state until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 195 mg: Subjects received 195 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 255 mg: Subjects received 255 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
ng/mL
  C1D1 | 1.65 (59.2) | 2.87 (56.6) | 4.55 (113.4) | 17.26 (27.8) | 30.90 (32.6) | 39.19 (69.7) | 187.98 (39.7) | 321.85 (32.7) | 306.63 (110.4) | 373.59 (24.9) | 605.11 (48.8) | 539.02 (78.0) | 680.87 (45.6) | 990.92 (64.9)
  C1D15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 11 | 4
  C1D15 | 2.28 (58.0) | 7.77 (96.2) | 4.21 (39.9) | 18.78 (32.2) | 18.47 (33.1) | 34.87 (36.8) | 131.71 (14.7) | 286.88 (21.8) | 539.17 (37.1) | 432.46 (7.6) | 492.81 (117.1) | 450.29 (67.4) | 629.85 (71.3) | 1535.60 (57.1)
  C3D1: number analyzed (Participants) | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 8 | 7 | 3
  C3D1 | 1.25 (5.7) | 4.30 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 6.56 (39.8) | 14.81 (50.1) | 16.10 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 96.60 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 710.94 (57.4) | 532.80 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 568.49 (76.2) | 795.86 (50.0) | 773.14 (51.0) | 2344.91 (23.1)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MSC1936369B: Regimen 2 (With Food Effect)
Description: Cmax was obtained directly from the concentration versus time curve. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: The food effect analysis set included all subjects who fulfilled following conditions: Food & drink intake, trial medication administration according to protocol, & not excreted irregularly, PK samples collected. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MSC1936369B 90 mg: Subjects received 90 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 and Day 2 of 21-day treatment cycle in either fed or fasted state until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
ng/mL
  Fasted | 321.14 (58.3) | 1158.00 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 305.94 (45.6) | 370.70 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MSC1936369B: Regimen 3 Once Daily
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies the subjects who were evaluated at that specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MSC1936369B 60 mg: Subjects received 60 mg of MSC1936369B (capsule formulation) orally, QD in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
ng/mL
  C1D1 | 241.27 (47.0) | 402.77 (59.2)
  C1D15 | 316.08 (34.9) | 324.80 (65.8)
  C3D1: number analyzed (Participants) | 2 | 10
  C3D1 | 473.27 (38.7) | 376.62 (45.2)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MSC1936369B: Regimen 3 Twice Daily
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, and 10 h post-dose on Cycle 1 Day 1 and Day 15; pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 h post dose on Cycle 3 Day 1
Population: PKS analysis set. Here "Number analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MSC1936369B 45 mg: Subjects received 45 mg of MSC1936369B (capsule formulation) orally, BID in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 60 mg: Subjects received 60 mg of MSC1936369B (capsule formulation) orally, BID in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 75 mg: Subjects received 75 mg of MSC1936369B (capsule formulation) orally, BID in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 18 | 13
ng/mL
  C1D1 | 132.57 (40.2) | 206.46 (41.7) | 263.08 (68.5)
  C1D15: number analyzed (Participants) | 3 | 18 | 11
  C1D15 | 178.09 (95.0) | 231.12 (44.0) | 190.42 (57.6)
  C3D1: number analyzed (Participants) | 2 | 13 | 6
  C3D1 | 139.60 (26.6) | 157.46 (53.7) | 329.28 (73.5)

10. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MSC1936369B: Regimen 1
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 4 | 3 | 13
Hours (h)
  C1D1 | 1.500 [1.02 to 1.53] | 0.750 [0.50 to 4.25] | 1.500 [1.00 to 2.50] | 1.500 [1.00 to 2.17] | 1.500 [1.00 to 2.50] | 1.000 [0.50 to 2.00] | 1.500 [1.00 to 4.00] | 1.017 [1.00 to 2.50] | 1.000 [0.98 to 1.50] | 1.483 [0.52 to 2.17] | 1.017 [0.50 to 6.00]
  C1D12: number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 11
  C1D12 | 1.633 [0.50 to 2.50] | 0.533 [0.33 to 2.00] | 1.000 [1.00 to 2.50] | 1.000 [1.00 to 1.08] | 1.017 [1.00 to 1.05] | 1.500 [1.50 to 1.50] | 1.000 [0.50 to 3.92] | 2.000 [0.75 to 2.52] | 1.000 [0.50 to 4.00] | 1.500 [1.50 to 2.00] | 1.083 [0.52 to 8.00]
  C3D1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 1 | 3 | 2 | 0 | 2 | 7
  C3D1 | 1.52 [1.52 to 1.52] | 0.500 [0.50 to 0.50] | 1.52 [1.52 to 1.52] | 1.000 [0.50 to 2.67] | 1.517 [1.00 to 4.05] | 1.500 [1.50 to 1.50] | 1.000 [1.00 to 3.58] | 1.508 [0.50 to 2.52] |  | 1.767 [1.50 to 2.03] | 2.000 [0.50 to 4.00]

11. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MSC1936369B: Regimen 2 (Without Food Effect)
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours (h)
Groups:
- MSC1936369B 3.5 mg: Subjects received 3.5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
- MSC1936369B 68 mg: Subjects received 68 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
Hours (h)
  C1D1 | 1.500 [1.50 to 1.92] | 1.017 [0.50 to 2.50] | 1.500 [1.00 to 2.00] | 1.000 [0.50 to 24.98] | 0.533 [0.52 to 2.00] | 1.500 [0.50 to 4.00] | 1.000 [0.58 to 2.02] | 0.500 [0.50 to 1.02] | 1.000 [0.47 to 1.50] | 1.500 [0.50 to 1.58] | 1.250 [0.33 to 2.02] | 1.500 [0.58 to 4.00] | 1.250 [0.50 to 2.50] | 2.000 [0.50 to 2.50]
  C1D15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 11 | 4
  C1D15 | 1.500 [1.42 to 2.00] | 0.967 [0.52 to 1.50] | 2.000 [0.43 to 2.00] | 0.667 [0.50 to 2.50] | 1.008 [1.00 to 1.02] | 1.500 [1.50 to 4.00] | 1.017 [0.50 to 2.12] | 1.500 [0.67 to 1.52] | 1.250 [1.00 to 1.50] | 1.500 [1.50 to 2.02] | 2.000 [1.00 to 2.08] | 1.517 [1.00 to 7.92] | 1.250 [0.50 to 3.00] | 1.458 [1.00 to 2.00]
  C3D1: number analyzed (Participants) | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 8 | 7 | 3
  C3D1 | 1.250 [1.00 to 1.50] | 2.000 [2.00 to 2.00] | 1.258 [1.00 to 1.52] | 1.000 [1.00 to 1.00] | 2.500 [2.50 to 2.50] |  | 1.50 [1.50 to 1.50] |  | 0.500 [0.50 to 0.50] | 2.000 [2.00 to 2.00] | 1.042 [0.58 to 1.50] | 1.333 [1.00 to 2.10] | 1.000 [0.50 to 2.02] | 1.000 [1.00 to 1.67]

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MSC1936369B: Regimen 2 (With Food Effect)
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: The food effect analysis set (FES). Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
Hours (h)
  Fasted | 1.600 [0.33 to 2.50] | 1.000 [1.00 to 1.00]
  Fed | 2.033 [1.50 to 4.00] | 6.000 [6.00 to 6.00]

13. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MSC1936369B: Regimen 3 Once Daily
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
Hours (h)
  C1D1 | 1.033 [1.00 to 1.50] | 1.500 [0.50 to 2.03]
  C1D15 | 2.500 [1.52 to 2.50] | 1.492 [0.50 to 4.00]
  C3D1: number analyzed (Participants) | 2 | 10
  C3D1 | 2.000 [1.50 to 2.50] | 1.000 [0.57 to 2.10]

14. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MSC1936369B: Regimen 3 Twice Daily
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 9
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 18 | 13
Hours (h)
  C1D1 | 1.500 [1.00 to 2.00] | 1.000 [0.50 to 4.00] | 0.667 [0.47 to 2.50]
  C1D15: number analyzed (Participants) | 3 | 18 | 11
  C1D15 | 1.500 [1.03 to 2.00] | 1.500 [0.50 to 2.55] | 1.500 [0.97 to 4.08]
  C3D1: number analyzed (Participants) | 2 | 13 | 6
  C3D1 | 1.467 [0.92 to 2.02] | 1.183 [0.50 to 2.07] | 1.467 [0.50 to 1.57]

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of MSC1936369B: Regimen 1
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- MSC1936369B 68 mg: Subjects received 68 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 4 | 3 | 13
hour*nanogram per milliliter (h*ng/mL)
  C1D1 | 4.6 (431.3) | 5.2 (63.9) | 18.5 (49.8) | 22.7 (29.2) | 52.7 (74.5) | 213.9 (84.0) | 531.3 (55.4) | 889.0 (31.9) | 1624.8 (36.1) | 1748.1 (38.8) | 2292.4 (52.5)
  C1D12: number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 11
  C1D12 | 7.0 (269.8) | 6.0 (89.3) | 26.0 (55.0) | 35.9 (79.7) | 83.6 (67.7) | 182.0 (125.1) | 691.9 (51.4) | 880.0 (45.7) | 1900.3 (99.7) | 1991.4 (19.2) | 1682.4 (52.4)
  C3D1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 1 | 3 | 2 | 0 | 2 | 7
  C3D1 | 6.9 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.7 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 21.0 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 23.0 (38.2) | 45.2 (51.8) | 113.2 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 334.9 (47.8) | 666.3 (52.3) |  | 876.7 (20.4) | 2064.1 (55.0)

16. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of MSC1936369B: : Regimen 2 (Without Food Effect)
Description: as for outcome 15
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure and "Number Analyzed" signifies those who were evaluated at the specified time point. Data was not available for categories with Number Analyzed=0 because there was no subject analyzed at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
hour*ng/mL
  C1D1 | 1.9 (331.6) | 8.2 (53.1) | 6.7 (292.9) | 67.9 (93.9) | 74.4 (19.4) | 188.4 (61.7) | 625.7 (20.6) | 808.0 (15.7) | 861.1 (112.4) | 1484.6 (13.0) | 2287.0 (96.6) | 2216.5 (75.7) | 3415.6 (44.5) | 4041.3 (60.8)
  C1D15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 11 | 4
  C1D15 | 4.3 (228.5) | 22.2 (42.1) | 13.8 (66.9) | 79.3 (57.9) | 67.8 (53.9) | 161.5 (14.1) | 621.2 (12.7) | 906.3 (15.4) | 1553.9 (122.5) | 1826.2 (17.9) | 1862.3 (96.4) | 2086.6 (69.9) | 3436.8 (64.7) | 5765.9 (15.3)
  C3D1: number analyzed (Participants) | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 8 | 7 | 3
  C3D1 | 0.5 (76.6) | 10.2 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 26.2 (15.6) | 40.5 (26.9) | 46.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 306.2 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 1394.7 (24.6) | 1299.3 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2053.6 (71.1) | 2171.2 (59.4) | 2484.5 (53.6) | 4906.3 (19.2)

17. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of MSC1936369B: Regimen 2 (With Food Effect)
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
hour*ng/mL
  Fasted | 1509.6 (46.6) | 3286 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 1458.3 (41.3) | 5072.9 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of MSC1936369B: Regimen 3 Once Daily
Description: as for outcome 15
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
hour*ng/mL
  C1D1 | 1229.3 (96.5) | 1544.9 (57.1)
  C1D15 | 1532.4 (80.4) | 1428.8 (63.6)
  C3D1: number analyzed (Participants) | 2 | 10
  C3D1 | 1392.3 (35.2) | 1122.5 (45.2)

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of MSC1936369B: Regimen 3 Twice Daily
Description: as for outcome 15
Time Frame: as for outcome 9
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 18 | 13
hour*ng/mL
  C1D1 | 407.2 (40.7) | 681.4 (43.7) | 791.1 (62.3)
  C1D15: number analyzed (Participants) | 3 | 18 | 11
  C1D15 | 589.3 (66.5) | 838.8 (43.9) | 710.3 (65.0)
  C3D1: number analyzed (Participants) | 2 | 13 | 6
  C3D1 | 450.0 (57.1) | 577.0 (72.5) | 1005.0 (25.6)

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MSC1936369B : Regimen 1
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 3 | 3 | 6 | 3 | 4 | 3 | 12
hour*ng/mL
  C1D1 | 136.2 (9.2) | 6.2 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 55.5 (321.8) | 31.4 (29.7) | 61.3 (66.9) | 234.1 (70.2) | 574.2 (50.0) | 924.2 (32.7) | 1699.7 (36.1) | 1836.4 (42.8) | 2773.5 (54.7)
  C1D12: number analyzed (Participants) | 2 | 1 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 9
  C1D12 | 38.3 (254.8) | 9.4 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 43.8 (58.7) | 47.5 (68.1) | 105.6 (57.6) | 206.3 (106.5) | 805.6 (58.9) | 960.7 (46.9) | 2108.2 (115.0) | 2257.6 (30.1) | 2022.8 (41.3)
  C3D1: number analyzed (Participants) | 1 | 0 | 1 | 3 | 2 | 1 | 2 | 2 | 0 | 2 | 6
  C3D1 | 15.4 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 47.6 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 34.4 (37.6) | 55.5 (90.0) | 134.5 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 489.8 (55.2) | 1072.1 (121.6) |  | 1056.0 (26.6) | 3477.6 (102.0)

21. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MSC1936369B: Regimen 2 (Without Food Effect)
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the Lower Limit of quantification (LLQ) and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
hour*ng/mL
  C1D1: number analyzed (Participants) | 0 | 2 | 2 | 2 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
  C1D1 |  | 23.4 (65.7) | 23.6 (22.5) | 59.1 (6.2) | 90.3 (30.8) | 218.4 (62.1) | 646.9 (20.7) | 820.4 (15.7) | 885.8 (111.0) | 1525.6 (13.2) | 2424.2 (109.7) | 2287.8 (77.4) | 3602.2 (46.2) | 4300.3 (54.2)
  C1D15: number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 8 | 10 | 4
  C1D15 | 15.7 (10.6) | 33.3 (45.8) | 21.9 (91.5) | 102.0 (63.6) | 89.7 (85.9) | 172.2 (9.0) | 669.1 (10.5) | 933.9 (15.4) | 1665.2 (132.1) | 1893.2 (17.5) | 2129.0 (123.7) | 2029.9 (63.3) | 3900.8 (64.3) | 6232.1 (7.0)
  C3D1: number analyzed (Participants) | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 8 | 7 | 3
  C3D1 |  | 15.4 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 41.2 (41.4) | 49.5 (17.4) | 58.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 415.6 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 1655.1 (19.1) | 1584.8 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2461.3 (64.3) | 2796.2 (59.3) | 3452.9 (61.6) | 5651.1 (23.5)

22. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MSC1936369B: Regimen 2 (With Food Effect)
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
hour*ng/mL
  Fasted | 1580.6 (48.7) | 3344.3 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 1495.7 (41.8) | 5633.8 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

23. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MSC1936369B: Regimen 3 Twice Daily
Description: as for outcome 20
Time Frame: as for outcome 9
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 18 | 13
hour*ng/mL
  C1D1: number analyzed (Participants) | 3 | 17 | 13
  C1D1 | 527.6 (57.4) | 742.3 (47.1) | 939.9 (67.3)
  C1D15: number analyzed (Participants) | 3 | 18 | 11
  C1D15 | 674.1 (73.6) | 1004.2 (46.4) | 978.4 (63.7)
  C3D1: number analyzed (Participants) | 2 | 13 | 6
  C3D1 | 696.0 (101.4) | 700.8 (79.0) | 1285.7 (29.0)

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MSC1936369B: Regimen 3 Once Daily
Description: as for outcome 20
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
hour*ng/mL
  C1D1 | 1253.1 (96.9) | 1581.4 (56.6)
  C1D15 | 1753.9 (93.1) | 1517.1 (65.6)
  C3D1: number analyzed (Participants) | 2 | 10
  C3D1 | 1597.0 (50.7) | 1400.3 (53.0)

25. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MSC1936369B: Regimen 1
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz. As AUCextra was >20% of AUC0-inf, t1/2 derived from λz was regarded as implausible & not calculated for arms MSC1936369B 1mg, 1.5mg, 2.5 mg.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 3 | 6 | 3 | 4 | 3 | 10
Hours (h)
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 3 | 6 | 3 | 4 | 3 | 10
  C1D1 |  |  |  | 3.346 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 3.405 (52.1) | 4.599 (29.1) | 4.781 (39.4) | 5.389 (9.4) | 5.335 (23.6) | 5.351 (15.9) | 5.247 (17.1)
  C1D12: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 3 | 4 | 3 | 3 | 2 | 8
  C1D12 |  |  |  | 4.985 (123.5) | 9.249 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 3.236 (19.4) | 6.750 (21.5) | 4.688 (60.4) | 6.926 (33.6) | 5.672 (15.4) | 3.964 (44.7)
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3
  C3D1 |  |  |  |  | 2.959 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.811 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 2.931 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 2.842 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 3.038 (3.4)

26. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MSC1936369B: Regimen 2 (Without Food Effect)
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz. As AUCextra was >20% of AUC0-inf, t1/2 derived from λz was regarded as implausible & not calculated for arms MSC1936369B 1mg, 2mg, 3.5 mg.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Groups:
- MSC1936369B 94 mg: Subjects received 94 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
Hours (h)
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
  C1D1 |  |  |  |  | 2.594 (5.0) | 5.119 (30.5) | 5.115 (6.6) | 4.187 (10.3) | 3.305 (84.0) | 4.826 (14.0) | 5.057 (45.3) | 4.904 (18.8) | 5.641 (21.6) | 4.313 (29.6)
  C1D15: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 7 | 10 | 4
  C1D15 |  |  |  | 2.941 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.335 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 4.443 (67.3) | 6.646 (19.5) | 5.277 (8.0) | 6.441 (28.4) | 5.193 (11.1) | 4.851 (7.9) | 5.479 (14.1) | 6.016 (18.9) | 4.847 (16.4)
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4 | 3 | 2
  C3D1 |  |  |  | 2.732 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  |  |  |  | 3.477 (11.0) | 2.853 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.863 (22.0) | 2.418 (25.2) | 2.628 (9.4) | 2.260 (34.4)

27. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MSC1936369B: Regimen 2 (With Food Effect)
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
Hour (h)
  Fasted | 4.898 (36.7) | 4.452 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 4.534 (18.3) | 6.123 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

28. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MSC1936369B: Regimen 3 Once Daily
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
Hour (h)
  C1D1 | 4.236 (1.3) | 4.097 (33.5)
  C1D15: number analyzed (Participants) | 2 | 12
  C1D15 | 5.259 (14.8) | 5.599 (30.1)
  C3D1: number analyzed (Participants) | 1 | 6
  C3D1 | 1.780 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.680 (21.1)

29. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MSC1936369B: Regimen 3 Twice Daily
Description: as for outcome 28
Time Frame: as for outcome 9
Population: PKS analysis set. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure and "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 17 | 12
Hour (h)
  C1D1: number analyzed (Participants) | 1 | 17 | 12
  C1D1 | 2.050 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.509 (25.1) | 2.814 (20.2)
  C1D15: number analyzed (Participants) | 3 | 14 | 7
  C1D15 | 2.890 (23.8) | 3.265 (18.6) | 3.210 (23.8)
  C3D1: number analyzed (Participants) | 1 | 7 | 2
  C3D1 | 3.144 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 2.636 (17.0) | 3.260 (10.6)

30. Secondary Outcome: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of MSC1936369B: Regimen 1
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from plasma, CL= Dose/AUC0-inf. As AUCextra was >20% of AUC0-inf, CL/f derived from λz was regarded as implausible & not calculated for arms MSC1936369B 1mg, 1.5mg, 2.5 mg.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 3 | 6 | 3 | 4 | 3 | 10
Liter per hour
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 3 | 6 | 3 | 4 | 3 | 10
  C1D1 |  |  |  | 132.69 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 114.26 (66.9) | 59.80 (70.2) | 48.76 (50.0) | 48.69 (32.7) | 40.01 (36.1) | 50.45 (41.2) | 47.82 (53.3)
  C1D12: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 3 | 4 | 3 | 3 | 2 | 8
  C1D12 |  |  |  | 70.60 (77.3) | 44.55 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 62.53 (92.6) | 37.49 (55.2) | 49.37 (43.8) | 35.80 (99.7) | 50.88 (19.6) | 61.44 (42.3)
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3
  C3D1 |  |  |  |  | 217.56 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 104.07 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 82.35 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 107.06 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 72.25 (35.7)

31. Secondary Outcome: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of MSC1936369B: Regimen 2 (Without Food Effect)
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from plasma, CL= Dose/AUC0-inf. As AUCextra was >20% of AUC0-inf, CL/f derived from λz was regarded as implausible & not calculated for arms MSC1936369B 1mg, 2mg, 3.5 mg.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
Liter per hour
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
  C1D1 |  |  |  |  | 90.76 (18.3) | 64.09 (62.1) | 43.28 (20.7) | 54.85 (15.7) | 76.77 (111.0) | 61.61 (13.2) | 49.50 (109.7) | 65.57 (77.4) | 54.13 (46.2) | 60.63 (53.4)
  C1D15: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 7 | 10 | 4
  C1D15 |  |  |  | 59.55 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 134.9 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 86.72 (12.5) | 45.10 (12.7) | 49.65 (15.4) | 43.76 (122.4) | 51.47 (17.9) | 92.42 (84.1) | 81.22 (65.4) | 53.49 (64.3) | 42.20 (5.9)
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4 | 3 | 2
  C3D1 |  |  |  | 89.34 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  |  |  |  | 41.08 (19.1) | 59.31 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 48.76 (64.3) | 61.04 (53.0) | 72.33 (63.8) | 44.23 (37.5)

32. Secondary Outcome: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of MSC1936369B: Regimen 2 (With Food Effect)
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from plasma, CL= Dose/AUC0-inf. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
Liter per hour
  Fasted | 56.94 (48.7) | 44.85 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 60.17 (41.8) | 26.62 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

33. Secondary Outcome: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of MSC1936369B: Regimen 3 Once Daily
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from plasma, CL= Dose/AUC0-inf.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
Liter per hour
  C1D1 | 47.88 (96.9) | 56.91 (56.6)
  C1D15: number analyzed (Participants) | 2 | 12
  C1D15 | 48.31 (103.9) | 62.85 (63.6)
  C3D1: number analyzed (Participants) | 1 | 6
  C3D1 | 53.36 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 75.63 (59.6)

34. Secondary Outcome: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of MSC1936369B: Regimen 3 Twice Daily
Description: as for outcome 33
Time Frame: as for outcome 9
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 17 | 12
Liter per hour
  C1D1: number analyzed (Participants) | 1 | 17 | 12
  C1D1 | 114.82 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 80.83 (47.1) | 83.86 (67.2)
  C1D15: number analyzed (Participants) | 3 | 14 | 7
  C1D15 | 71.44 (69.3) | 66.89 (52.1) | 94.48 (71.2)
  C3D1: number analyzed (Participants) | 1 | 7 | 2
  C3D1 | 126.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 103.3 (66.9) | 77.09 (21.0)

35. Secondary Outcome: Apparent Volume of Distribution Following Extravascular Administration (Vz/F) of MSC1936369B: Regimen 1
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by λz. As AUCextra was >20% of AUC0-inf, Vz/F derived from λz was regarded as implausible & not calculated for arms MSC1936369B 1mg, 1.5mg, 2.5 mg.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Groups:
- MSC1936369B 3.5 mg: Subjects received 3.5 mg of MSC1936369B (capsule formulation) orally, QD on Days 1 to 5, 8 to 12, 15 to 19 of each 21-day treatment cycle.
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 3 | 6 | 3 | 4 | 3 | 10
Liter
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 3 | 6 | 3 | 4 | 3 | 10
  C1D1 |  |  |  | 640.60 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 561.27 (12.9) | 396.76 (86.7) | 336.32 (78.8) | 378.56 (23.0) | 307.90 (43.1) | 389.49 (28.6) | 361.99 (43.0)
  C1D12: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 3 | 4 | 3 | 3 | 2 | 8
  C1D12 |  |  |  | 507.8 (28.3) | 594.5 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 291.9 (73.0) | 365.1 (35.0) | 333.9 (65.1) | 357.8 (53.7) | 416.3 (35.8) | 351.4 (37.5)
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3
  C3D1 |  |  |  |  | 928.91 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 422.04 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 348.19 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 438.91 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 316.63 (33.9)

36. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Following Extravascular Administration (Vz/F) of MSC1936369B: Regimen 2 (Without Food Effect)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by λz. As AUCextra was >20% of AUC0-inf, Vz/F derived from λz was regarded as implausible & not calculated for arms MSC1936369B 1mg, 2mg, 3.5 mg.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
Liter
  C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
  C1D1 |  |  |  |  | 339.58 (13.2) | 473.32 (81.2) | 319.40 (27.0) | 331.36 (13.3) | 366.00 (22.8) | 428.99 (22.7) | 361.12 (58.1) | 463.92 (68.7) | 440.55 (41.7) | 377.28 (42.4)
  C1D15: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 7 | 10 | 4
  C1D15 |  |  |  | 252.7 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 454.6 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 555.9 (84.7) | 432.5 (30.7) | 378.0 (23.6) | 406.6 (76.5) | 385.6 (25.9) | 646.9 (96.3) | 642.1 (63.5) | 464.2 (64.9) | 295.1 (13.4)
  C3D1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4 | 3 | 2
  C3D1 |  |  |  | 352.10 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  |  |  |  | 206.07 (30.5) | 244.16 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 201.39 (95.6) | 212.92 (34.4) | 274.24 (53.8) | 144.24 (79.1)

37. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Following Extravascular Administration (Vz/F) of MSC1936369B: Regimen 2 (With Food Effect)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by λz. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: The food effect analysis set (FES). Here, "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome Measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
Liter
  Fasted | 402.4 (49.0) | 288.1 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 393.6 (40.5) | 235.2 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

38. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Following Extravascular Administration (Vz/F) of MSC1936369B: Regimen 3 Once Daily
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by λz
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
Liter
  C1D1 | 292.61 (99.0) | 336.38 (47.1)
  C1D15: number analyzed (Participants) | 2 | 12
  C1D15 | 366.5 (131.6) | 507.7 (66.0)
  C3D1: number analyzed (Participants) | 1 | 6
  C3D1 | 137.0 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 292.5 (47.3)

39. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Following Extravascular Administration (Vz/F) of MSC1936369B: Regimen 3 Twice Daily
Description: as for outcome 38
Time Frame: as for outcome 9
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 17 | 12
Liter
  C1D1: number analyzed (Participants) | 1 | 17 | 12
  C1D1 | 339.51 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 292.59 (42.3) | 340.43 (57.7)
  C1D15: number analyzed (Participants) | 3 | 14 | 7
  C1D15 | 297.9 (57.8) | 315.0 (59.4) | 437.6 (59.1)
  C3D1: number analyzed (Participants) | 1 | 7 | 2
  C3D1 | 571.8 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 392.9 (81.9) | 362.6 (10.2)

40. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated From Last Observation to Infinity Given as Percentage of AUC 0-∞ (AUC Extra): Regimen 1
Description: AUCextra was defined as a percentage of AUC0-inf obtained by extrapolation: %AUCextra = (1- [AUC0-t / AUC0-inf])*100. %AUCextra was reported in terms of percentage of AUC0-inf.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 12 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC 0-∞
Arm/Group | MSC1936369B 1 mg | MSC1936369B 1.5 mg | MSC1936369B 2.5 mg | MSC1936369B 3.5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 3 | 3 | 6 | 3 | 4 | 3 | 12
Percentage of AUC 0-∞
  C1D1 | 81.33 (21.2) | 42.23 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 43.45 (79.8) | 26.80 (27.3) | 13.08 (47.7) | 5.31 (174.3) | 5.39 (112.5) | 3.52 (52.0) | 4.08 (47.3) | 4.09 (75.2) | 5.28 (155.8)
  C1D12: number analyzed (Participants) | 2 | 1 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 9
  C1D12 | 50.60 (8.6) | 33.84 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 40.60 (5.6) | 21.27 (56.8) | 19.82 (37.6) | 7.83 (193.6) | 6.57 (45.0) | 8.17 (29.1) | 6.56 (185.5) | 7.94 (131.8) | 2.97 (137.2)
  C3D1: number analyzed (Participants) | 1 | 0 | 1 | 3 | 2 | 1 | 2 | 2 | 0 | 2 | 6
  C3D1 | 55.15 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 55.79 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 32.85 (14.3) | 21.27 (33.1) | 15.84 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 28.06 (30.6) | 27.67 (126.0) |  | 16.54 (30.2) | 26.05 (98.7)

41. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated From Last Observation to Infinity Given as Percentage of AUC 0-∞ (AUC Extra): Regimen 2 (Without Food Effect)
Description: as for outcome 40
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC 0-∞
Arm/Group | MSC1936369B 1 mg | MSC1936369B 2 mg | MSC1936369B 3.5 mg | MSC1936369B 5 mg | MSC1936369B 7 mg | MSC1936369B 14 mg | MSC1936369B 28 mg | MSC1936369B 45 mg | MSC1936369B 68 mg | MSC1936369B 94 mg | MSC1936369B 120 mg | MSC1936369B 150 mg | MSC1936369B 195 mg | MSC1936369B 255 mg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
Percentage of AUC 0-∞
  C1D1: number analyzed (Participants) | 0 | 2 | 2 | 2 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 14 | 12 | 5
  C1D1 |  | 55.78 (11.0) | 31.63 (31.2) | 27.25 (15.2) | 15.10 (63.9) | 12.17 (59.8) | 3.29 (3.7) | 1.46 (30.8) | 2.66 (40.8) | 2.60 (33.4) | 2.94 (181.0) | 2.64 (68.3) | 4.36 (76.2) | 3.57 (149.3)
  C1D15: number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 8 | 10 | 4
  C1D15 | 40.86 (2.9) | 33.34 (6.4) | 35.29 (30.0) | 21.93 (20.2) | 19.45 (107.4) | 12.45 (58.0) | 6.89 (32.9) | 2.96 (1.9) | 5.00 (141.4) | 3.40 (33.9) | 5.82 (251.8) | 4.82 (82.9) | 5.77 (72.8) | 5.22 (112.2)
  C3D1: number analyzed (Participants) | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 8 | 7 | 3
  C3D1 |  | 33.93 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 33.77 (47.7) | 17.27 (45.0) | 20.68 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 26.32 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. |  | 15.35 (29.7) | 18.02 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group. | 16.22 (26.9) | 17.54 (83.4) | 23.45 (59.4) | 11.15 (77.4)

42. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated From Last Observation to Infinity Given as Percentage of AUC 0-∞ (AUC Extra): Regimen 2 (With Food Effect)
Description: AUCextra was defined as a percentage of AUC0-inf obtained by extrapolation: AUCextra = (1- [AUC0-t / AUC0-inf])*100. AUCextra was reported in terms of percentage of AUC0-inf. Summarized data over Day 1 and Day 2 was reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12 and 24 hours post-dose on Cycle 1 Day 1 and Day 2
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC 0-∞
Arm/Group | MSC1936369B 90 mg | MSC1936369B 150 mg
Number analyzed (Participants) | 8 | 1
Percentage of AUC 0-∞
  Fasted | 2.54 (149.8) | 1.74 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.
  Fed | 2.21 (56.3) | 9.96 (NA) — Geometric Coefficient of Variation could not be calculated as there was only 1 subject analyzed in this reporting group.

43. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated From Last Observation to Infinity Given as Percentage of AUC 0-∞ (AUC Extra): Regimen 3 Once Daily
Description: AUCextra was defined as a percentage of AUC0-inf obtained by extrapolation: AUCextra = (1- [AUC0-t / AUC0-inf])*100. AUCextra was reported in terms of percentage of AUC0-inf.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 3 Day 1
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC 0-∞
Arm/Group | MSC1936369B 60 mg | MSC1936369B 90 mg
Number analyzed (Participants) | 3 | 12
percentage of AUC 0-∞
  C1D1 | 1.88 (16.2) | 2.11 (50.0)
  C1D15 | 7.95 (149.3) | 4.28 (85.0)
  C3D1: number analyzed (Participants) | 2 | 10
  C3D1 | 9.11 (171.3) | 17.56 (50.9)

44. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated From Last Observation to Infinity Given as Percentage of AUC 0-∞ (AUC Extra): Regimen 3 Twice Daily
Description: as for outcome 43
Time Frame: as for outcome 9
Population: PKS analysis set. Here "Number Analyzed" signifies those who were evaluated at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC 0-∞
Arm/Group | MSC1936369B 45 mg | MSC1936369B 60 mg | MSC1936369B 75 mg
Number analyzed (Participants) | 3 | 18 | 13
Percentage of AUC 0-∞
  C1D1: number analyzed (Participants) | 3 | 17 | 13
  C1D1 | 16.82 (128.4) | 7.70 (58.3) | 10.90 (68.3)
  C1D15: number analyzed (Participants) | 3 | 18 | 11
  C1D15 | 11.78 (42.8) | 14.14 (51.4) | 19.19 (79.3)
  C3D1: number analyzed (Participants) | 2 | 13 | 6
  C3D1 | 30.63 (70.7) | 16.43 (37.5) | 21.34 (21.8)

45. Secondary Outcome: Phosphorylated Extra-Cellular Signal-Regulated Kinase (pERK) Fold Change in Peripheral Blood Monocyte Cells (PBMC) and Tot ERK Fold Change in Peripheral Blood Monocyte Cells (PBMC)
Time Frame: Pre-dose on C1D1, C1D2, C1D5, C1D8; 2, 4, 8 h post-dose on C1D1; pre-dose, 2, 8, 24 h post-dose on C1D12-15; pre-dose, 2, 4 h post-dose on C1D3
Population: Analysis population included subjects from safety analysis set having at least one pERK/tot ERK sample and not excluded from the analysis as per SAP. Number analyzed= subjects who were evaluated at the specified time point. Data was not available for categories with Number analyzed=0 because there was no subject analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: fold change
Groups:
- MSC1936369B Regimen 3 Once Daily: Subjects received MSC1936369B capsules 60 or 90 mg orally QD in each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision.
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily | MSC1936369B Regimen 3 Twice Daily
Number analyzed (Participants) | 41 | 76 | 12 | 31
fold change
  C1D1, Pre-dose (pERK) | 4.524 (1.839) | 3.937 (1.662) | 4.121 (1.743) | 3.629 (1.491)
  C1D1, 2 h post-dose (pERK): number analyzed (Participants) | 30 | 63 | 12 | 30
  C1D1, 2 h post-dose (pERK) | 1.235 (0.295) | 1.305 (0.755) | 1.178 (0.194) | 1.249 (0.219)
  C1D1, 4 h post-dose (pERK): number analyzed (Participants) | 11 | 13 | 0 | 0
  C1D1, 4 h post-dose (pERK) | 3.828 (1.715) | 3.422 (1.902) |  |
  C1D1, 8 h post-dose (pERK): number analyzed (Participants) | 9 | 39 | 12 | 31
  C1D1, 8 h post-dose (pERK) | 1.454 (0.515) | 1.454 (0.403) | 1.878 (0.836) | 1.821 (0.514)
  C1D2, Pre-dose (pERK): number analyzed (Participants) | 9 | 40 | 12 | 25
  C1D2, Pre-dose (pERK) | 2.853 (1.399) | 2.411 (1.031) | 3.081 (1.249) | 2.069 (0.748)
  C1D5, Pre-dose (pERK): number analyzed (Participants) | 8 | 0 | 0 | 0
  C1D5, Pre-dose (pERK) | 2.722 (1.326) |  |  |
  C1D8, Pre-dose (pERK): number analyzed (Participants) | 36 | 69 | 12 | 28
  C1D8, Pre-dose (pERK) | 4.48 (2.119) | 2.868 (1.473) | 2.541 (1.338) | 2.235 (0.739)
  C1D12-15, Pre-dose (pERK): number analyzed (Participants) | 37 | 68 | 12 | 28
  C1D12-15, Pre-dose (pERK) | 3.257 (1.671) | 3.265 (1.845) | 3.241 (2.249) | 2.16 (0.814)
  C1D12-15, 2 h Post-dose (pERK): number analyzed (Participants) | 8 | 35 | 12 | 29
  C1D12-15, 2 h Post-dose (pERK) | 1.252 (0.217) | 1.293 (0.447) | 1.471 (0.529) | 1.315 (0.218)
  C1D12-15, 8 h Post-dose (pERK): number analyzed (Participants) | 8 | 35 | 12 | 29
  C1D12-15, 8 h Post-dose (pERK) | 1.514 (0.391) | 1.653 (0.571) | 1.902 (0.87) | 1.98 (0.827)
  C1D12-15, 24 h Post-dose (pERK): number analyzed (Participants) | 6 | 31 | 12 | 20
  C1D12-15, 24 h Post-dose (pERK) | 2.768 (1.594) | 2.476 (0.958) | 2.598 (1.185) | 2.043 (0.76)
  C3D1, Pre-dose (pERK): number analyzed (Participants) | 16 | 13 | 0 | 0
  C3D1, Pre-dose (pERK) | 5.179 (2.151) | 3.716 (1.875) |  |
  C3D1, 2 h Post-dose (pERK): number analyzed (Participants) | 12 | 4 | 0 | 0
  C3D1, 2 h Post-dose (pERK) | 1.795 (0.687) | 1.288 (0.327) |  |
  C3D1, 4 h Post-dose (pERK): number analyzed (Participants) | 4 | 9 | 0 | 0
  C3D1, 4 h Post-dose (pERK) | 3.106 (0.461) | 2.688 (2.065) |  |
  C1D1, Pre-dose (Tot ERK): number analyzed (Participants) | 40 | 74 | 12 | 31
  C1D1, Pre-dose (Tot ERK) | 1.1 (0.468) | 1.075 (0.25) | 1.02 (0.169) | 1.086 (0.277)
  C1D1, 2 h post-dose (Tot ERK): number analyzed (Participants) | 30 | 61 | 12 | 30
  C1D1, 2 h post-dose (Tot ERK) | 1.063 (0.215) | 1.069 (0.247) | 1.078 (0.151) | 1.079 (0.193)
  C1D1, 4 h post-dose (Tot ERK): number analyzed (Participants) | 11 | 13 | 0 | 0
  C1D1, 4 h post-dose (Tot ERK) | 1.059 (0.621) | 1.012 (0.286) |  |
  C1D1, 8 h post-dose (Tot ERK): number analyzed (Participants) | 9 | 37 | 12 | 31
  C1D1, 8 h post-dose (Tot ERK) | 1.058 (0.16) | 1.095 (0.31) | 1.078 (0.143) | 1.098 (0.161)
  C1D2, Pre-dose (Tot ERK): number analyzed (Participants) | 9 | 38 | 12 | 25
  C1D2, Pre-dose (Tot ERK) | 1.075 (0.103) | 1.13 (0.455) | 1.013 (0.273) | 1.108 (0.154)
  C1D5, Pre-dose (Tot ERK): number analyzed (Participants) | 8 | 0 | 0 | 0
  C1D5, Pre-dose (Tot ERK) | 1.163 (0.146) |  |  |
  C1D8, Pre-dose (Tot ERK): number analyzed (Participants) | 36 | 67 | 12 | 28
  C1D8, Pre-dose (Tot ERK) | 1.233 (0.674) | 1.108 (0.353) | 0.944 (0.117) | 1.049 (0.133)
  C1D12-15, Pre-dose (Tot ERK): number analyzed (Participants) | 37 | 66 | 12 | 28
  C1D12-15, Pre-dose (Tot ERK) | 1.223 (0.476) | 1.118 (0.268) | 1.333 (0.878) | 1.047 (0.144)
  C1D12-15, 2 h Post-dose (Tot ERK): number analyzed (Participants) | 8 | 33 | 12 | 29
  C1D12-15, 2 h Post-dose (Tot ERK) | 1.04 (0.102) | 1.125 (0.34) | 1.335 (0.754) | 1.059 (0.14)
  C1D12-15, 8 h Post-dose (Tot ERK): number analyzed (Participants) | 8 | 33 | 12 | 29
  C1D12-15, 8 h Post-dose (Tot ERK) | 0.994 (0.165) | 1.041 (0.237) | 1.044 (0.238) | 1.026 (0.146)
  C1D12-15, 24 h Post-dose (Tot ERK): number analyzed (Participants) | 6 | 29 | 12 | 20
  C1D12-15, 24 h Post-dose (Tot ERK) | 1.047 (0.153) | 1.045 (0.183) | 1.048 (0.139) | 1.068 (0.141)
  C3D1, Pre-dose (Tot ERK): number analyzed (Participants) | 16 | 13 | 0 | 0
  C3D1, Pre-dose (Tot ERK) | 1.074 (0.34) | 1.138 (0.306) |  |
  C3D1, 2 h Post-dose (Tot ERK): number analyzed (Participants) | 12 | 4 | 0 | 0
  C3D1, 2 h Post-dose (Tot ERK) | 1.087 (0.413) | 1.251 (0.29) |  |
  C3D1, 4 h Post-dose (Tot ERK): number analyzed (Participants) | 4 | 9 | 0 | 0
  C3D1, 4 h Post-dose (Tot ERK) | 0.674 (0.304) | 1.052 (0.182) |  |

46. Secondary Outcome: Number of Subjects With Clinical Benefit (Complete Response [CR], Partial Response [PR] or Stable Disease [SD}) and Progressive Disease (PD) Based on the Best Overall Response (BOR)
Description: Number of subjects with clinical benefit (CR, PR, or SD) and PD according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0) was reported. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: defined as at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD:defined as at least a 20% increase in sum of longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of longest diameter while on study.
Time Frame: Baseline until disease progression (assessed up to end of treatment [253 weeks])
Population: The SAF included all subjects who received at least 1 administration of MSC1936369B. Here "Number of Subjects analysed" = subjects evaluable for this endpoint.
Measure: Number; unit: Subjects
Groups:
- MSC1936369B Regimen 2 and Regimen 2 Food Effect: Combined data for both Regimen 2 with and without food effect was reported in this arm. MSC1936369B Regimen 2: Subjects received MSC1936369B capsules 1 to 255 mg orally QD on Days 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision. MSC1936369B Regimen 2 (FE): Subjects received MSC1936369B capsules 90-150 mg orally QD on Day 1 to 15 of each 21-day treatment cycle until PD or intolerable toxicity or investigator/subject decision. Subjects in the Regimen 2 FE cohort were assigned either the fed/fasted sequence or fasted/fed sequence for Day 1 of Cycle 1 and Cycle 2 dosing.
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 and Regimen 2 Food Effect | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily
Number analyzed (Participants) | 39 | 71 | 15 | 33
Subjects
  CR | 0 | 0 | 0 | 1
  PR | 0 | 4 | 2 | 6
  SD | 19 | 34 | 9 | 14
  PD | 20 | 33 | 4 | 12

ADVERSE EVENTS:
Time Frame: Baseline up to 253 weeks
Description: The safety analysis set (SAF) included all subjects who received at least 1 administration of MSC1936369B.
Arm/Group | MSC1936369B Regimen 1 | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) | MSC1936369B Regimen 3 Once Daily (QD) | MSC1936369B Regimen 3 Twice Daily
Serious Adverse Events (participants affected / at risk) | 23/49 | 45/82 | 8/15 | 21/34
Other Adverse Events (participants affected / at risk) | 47/49 | 80/82 | 15/15 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSC1936369B Regimen 1 (N=49) | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) (N=82) | MSC1936369B Regimen 3 Once Daily (QD) (N=15) | MSC1936369B Regimen 3 Twice Daily (N=34)
General physical health deterioration (General disorders) | 7 | 13 | 2 | 2
Pyrexia (General disorders) | 2 | 3 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 4 | 0 | 1
Disease progression (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0
Obstruction (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Device occlusion (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 2 | 0 | 0 | 0
Choroiditis (Eye disorders) | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 2 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0
Macular oedema (Eye disorders) | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 2
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypoventilation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Macular detachment (Eye disorders) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSC1936369B Regimen 1 (N=49) | MSC1936369B Regimen 2 (Without Food Effect + With Food Effect) (N=82) | MSC1936369B Regimen 3 Once Daily (QD) (N=15) | MSC1936369B Regimen 3 Twice Daily (N=34)
Hypertension (Vascular disorders) | 7 | 4 | 1 | 4
Hot flush (Vascular disorders) | 4 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 1 | 2 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 2 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0
Vascular compression (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 27 | 38 | 8 | 12
Oedema peripheral (General disorders) | 12 | 30 | 9 | 21
Pyrexia (General disorders) | 9 | 13 | 3 | 12
Fatigue (General disorders) | 6 | 16 | 2 | 8
Non-cardiac chest pain (General disorders) | 2 | 3 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 1
Chills (General disorders) | 1 | 1 | 0 | 4
Hyperthermia (General disorders) | 1 | 1 | 0 | 1
Inflammation (General disorders) | 1 | 2 | 0 | 0
Influenza like illness (General disorders) | 1 | 2 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 2 | 3
Nodule (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 3 | 0 | 0
Face oedema (General disorders) | 0 | 3 | 1 | 8
Generalised oedema (General disorders) | 0 | 1 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 0 | 0
Mucosal dryness (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Thrombosis in device (General disorders) | 0 | 0 | 1 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 4
General physical health deterioration (General disorders) | 0 | 0 | 0 | 2
Localised oedema (General disorders) | 0 | 0 | 0 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 1
Injection site oedema (General disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 4 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 6 | 1 | 4
Anxiety (Psychiatric disorders) | 0 | 7 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 3 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Illusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Burn of internal organs (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Burn oesophageal (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 6 | 8 | 4 | 2
Ejection fraction decreased (Investigations) | 3 | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 1 | 5
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 2
Blood 25-hydroxycholecalciferol decreased (Investigations) | 1 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1
Blood parathyroid hormone increased (Investigations) | 1 | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram qt prolonged (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 2 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 3 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram pr prolongation (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Retinogram abnormal (Investigations) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 2 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 2
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 0 | 0
Colour blindness (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 10 | 22 | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 3 | 6 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6 | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 12 | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 3 | 7 | 1 | 5
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 5
Headache (Nervous system disorders) | 2 | 12 | 1 | 4
Somnolence (Nervous system disorders) | 2 | 3 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 0 | 2
Sciatica (Nervous system disorders) | 1 | 4 | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Viith nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 2
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 7 | 20 | 2 | 6
Visual impairment (Eye disorders) | 5 | 4 | 1 | 1
Colour blindness acquired (Eye disorders) | 4 | 1 | 0 | 0
Macular detachment (Eye disorders) | 3 | 14 | 9 | 16
Retinal detachment (Eye disorders) | 3 | 11 | 3 | 10
Eyelid oedema (Eye disorders) | 2 | 5 | 2 | 6
Photopsia (Eye disorders) | 2 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 2 | 1 | 1 | 1
Visual acuity reduced (Eye disorders) | 2 | 5 | 2 | 1
Altered visual depth perception (Eye disorders) | 1 | 0 | 0 | 0
Chromatopsia (Eye disorders) | 1 | 2 | 0 | 1
Corneal epithelium defect (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 3 | 0 | 0
Macular oedema (Eye disorders) | 1 | 1 | 0 | 1
Metamorphopsia (Eye disorders) | 1 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 3 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 2 | 0 | 0
Keratitis (Eye disorders) | 0 | 2 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 2 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Choroidal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1 | 0 | 3
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0
Growth of eyelashes (Eye disorders) | 0 | 1 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 1 | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 2 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 2 | 4
Eyelash discolouration (Eye disorders) | 0 | 0 | 1 | 0
Maculopathy (Eye disorders) | 0 | 0 | 1 | 0
Trichomegaly (Eye disorders) | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 1 | 0 | 3
Dry eye (Eye disorders) | 0 | 0 | 0 | 2
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 1
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 5 | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 25 | 46 | 14 | 29
Nausea (Gastrointestinal disorders) | 21 | 26 | 6 | 15
Vomiting (Gastrointestinal disorders) | 15 | 28 | 2 | 11
Stomatitis (Gastrointestinal disorders) | 10 | 12 | 1 | 8
Abdominal pain (Gastrointestinal disorders) | 9 | 17 | 1 | 10
Constipation (Gastrointestinal disorders) | 9 | 17 | 5 | 9
Dry mouth (Gastrointestinal disorders) | 6 | 6 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 7 | 0 | 6
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 2 | 2
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 4 | 2 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Aptyalism (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 9 | 13 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 18 | 6 | 14
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 19 | 7 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 9 | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 13 | 6 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 4 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 5
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 9 | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 7 | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 11 | 2 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 10 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 4 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 7 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 10 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 3 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 1
Erysipelas (Infections and infestations) | 1 | 1 | 1 | 2
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 2
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 2 | 2 | 5
Pharyngitis (Infections and infestations) | 1 | 4 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 5 | 1 | 5
Herpes virus infection (Infections and infestations) | 0 | 2 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 2 | 0 | 0
Anal infection (Infections and infestations) | 0 | 1 | 0 | 0
Chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 2
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 2
Eye infection (Infections and infestations) | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other